CLINICAL TRIAL: NCT04772612
Title: A Phase 1, Multicenter, Open-Label Study to Evaluate the Effect of Mild, Moderate, and Severe Hepatic Impairment on the Single-Dose Pharmacokinetics of Sitravatinib
Brief Title: A Study to Evaluate the Effect of Mild, Moderate, and Severe Hepatic Impairment on Pharmacokinetics of Sitravatinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 516-012
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — sitravatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sitravatinib in healthy subjects (Experimental): Participants will receive a single dose of sitravatinib 100 mg receive on Day 1 in healthy subjects.
  Interventions: Drug: sitravatinib
- Sitravatinib in subjects with mild hepatic impairment (Experimental): Participants will receive a single dose of sitravatinib 100 mg receive on Day 1 in subjects with mild hepatic impairment
  Interventions: Drug: sitravatinib
- Sitravatinib in subjects with moderate hepatic impairment (Experimental): Participants will receive a single dose of sitravatinib 100 mg receive on Day 1 in subjects with moderate hepatic impairment
  Interventions: Drug: sitravatinib
- Sitravatinib in subjects with severe hepatic impairment (Experimental): Participants will receive a single dose of sitravatinib 100 mg receive on Day 1 in subjects with severe hepatic impairment
  Interventions: Drug: sitravatinib

INTERVENTIONS:
Drug: sitravatinib — sitravatinib

SUMMARY:
A Phase 1, Multicenter, Open-Label Study to Evaluate the Effect of Mild, Moderate, and Severe Hepatic Impairment on the Single-Dose Pharmacokinetics of Sitravatinib

ELIGIBILITY:
Key Inclusion Criteria:

* Males or females, of any race, between 18 and 75 years of age, inclusive, at screening.
* Body mass index between 18.0 and 40.0 kg/m2, inclusive, at screening.
* Females of childbearing potential will not be pregnant or lactating and must have a negative result on an approved pregnancy test at screening and check-in. Females of childbearing potential must agree to use contraception by a method of proven reliability (including abstinence) as detailed in the protocol.
* Male subjects must agree to use contraception as detailed in the protocol.
* Able to comprehend and willing to sign an ICF and to abide by the study restrictions.

Participants with normal hepatic function must also satisfy the following criteria:

- Participants with normal hepatic function must be in good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, or clinical laboratory evaluations at screening and check-in as assessed by the investigator.

Participants with hepatic impairment must also satisfy the following criteria:

- Participants must meet the criteria for mild, moderate, or severe hepatic impairment based on Child Pugh (CP) score and classification as detailed in the protocol. Hepatically-impaired participants will be assigned to groups according to CP scores calculated at screening; CP scores will be recalculated at check-in to confirm that subjects do not have significant changes in status to ensure subject safety for the study, as determined by the investigator and medical monitor.

Key Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator.
* History of intestinal disease, inflammatory bowel disease, major gastric surgery, or other gastrointestinal conditions (eg, uncontrolled nausea, vomiting, malabsorption syndrome) likely to alter absorption of study treatment or result in inability to swallow oral medications (Cholecystectomy is not allowed.).
* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days or 5 half-lives prior to dosing, whichever is longer.
* Participants who, in the opinion of the investigator, should not participate in this study.

Participants with normal hepatic function will be excluded from the study if any of the following criteria are applicable:

* Significant history or clinical manifestation of any hepatic disease, as determined by lab abnormalities: AST, ALT, alkaline phosphatase, or alpha-fetoprotein >1 × upper limit of normal or as deemed clinically significant by the investigator.
* Participant has creatinine clearance <80 mL/minute as calculated by using the Cockcroft-Gault equation.
* Use or intend to use any prescription medications/products within 14 days prior to dosing, unless deemed acceptable by the investigator, medical monitor, and sponsor.

Participants with hepatic impairment will be excluded from the study if any of the following criteria are applicable:

* Ventricular dysfunction or history of risk factors for Torsades de Pointes (eg, unexplained syncope, known long QT syndrome, heart failure, and cardiomyopathy).
* Participant has had a change in disease status within 90 days prior to the study drug administration on Day 1, as documented by the subject's medical history, deemed clinically significant by the investigator.
* Participant has required a new medication or a change in medication dose within 2 weeks before dosing with sitravatinib.
* Participant has a current functioning organ transplant or is waiting for an organ transplant.
* History of unstable diabetes mellitus as evidenced by hemoglobin A1c ≥9% at screening.
* Uncontrolled arterial hypertension (> 150 mm Hg systolic or >100 mm Hg diastolic) on multiple observations despite standard of care treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - AUClast (sitravatinib) | 9 days
  AUC from time zero to the last measured time point
Pharmacokinetics - Tmax (sitravatinib) | 9 days
  Time to reach maximum observed plasma concentration
Pharmacokinetics - AUC∞ (sitravatinib) | 9 days
  Area under the plasma concentration-time curve from time zero extrapolated to infinity moderate, or severe hepatic impairment compared to control subjects with normal hepatic function
Pharmacokinetics - Cmax (sitravatinib) | 9 days
  Maximum observed plasma concentration
Pharmacokinetics - t1/2 (sitravatinib) | 9 days
  Terminal elimination half-life
Pharmacokinetics - CL/F (sitravatinib) | 9 days
  Apparent total plasma clearance when dosed orally
Pharmacokinetics - Vz/F (sitravatinib) | 9 days
  Apparent volume of distribution when dosed orally
Pharmacokinetics - fu (sitravatinib) | days 1 - 4
  Unbound fraction

SECONDARY OUTCOMES:
Adverse Events (AEs) | From the time the ICF is signed until 14 ± 2 days after the last dose of sitravatinib treatment
  Incidence and severity of adverse events (AEs).

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Chin, MD, Study Director — Mirati Therapeutics
Locations (5):
- United States (5):
  - Orange County Research Center, Tustin, California
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Nucleus Network, Saint Paul, Minnesota
  - Texas Liver Institute, Austin, Texas